CLINICAL TRIAL: NCT07152457
Title: Emergency Room Analgesia and Sedation Survey-2
Acronym: EASY-2
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0530; No funding is currently availa (Other: No funding is currently available.)
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Current Status of Analgesia and Sedation Cognition and Implementation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — None intervention

SUMMARY:
Part 1: Assessment of Healthcare Providers' Knowledge on Analgesia and Sedation in Emergency Resuscitation Rooms Across China This study aims to evaluate the understanding of healthcare providers in emergency resuscitation rooms regarding the principles of analgesia and sedation, commonly used assessment tools, and delirium management, and to identify key factors that may influence their level of knowledge. Part 2: Implementation Practices of Analgesia and Sedation in Emergency Resuscitation Rooms Across China: A Multicenter Prospective Cohort Study Primary Objective: To assess the extent of adherence to standardized protocols for analgesia and sedation in emergency resuscitation rooms of general hospitals in China. Secondary Objectives: (1) To identify key factors affecting compliance with standardized analgesia and sedation practices in emergency resuscitation settings, thereby providing evidence for targeted interventions; (2) To examine the impact of analgesia and sedation implementation on clinical outcomes and prognosis of patients in emergency resuscitation rooms.

ELIGIBILITY:
Inclusion Criteria:

1. ： Part 1: (1) Healthcare professionals currently assigned to the emergency department and actively working in the emergency resuscitation room; (2) With at least one year of clinical experience in emergency medicine; (3) Willing to voluntarily participate in the investigation. Each participating institution is required to enroll a minimum of 12 healthcare providers, including at least 6 physicians and 6 nurses. Within each group (physicians and nurses), at least 3 participants must hold junior professional titles and at least 3 must hold intermediate or senior-level professional titles.
2. Part 2: All adult patients (≥18 years of age) admitted to the emergency resuscitation room during the period from July 15, 2025 to July 30, 2025.

Exclusion Criteria:

1. Pregnant women
2. patients undergoing end-of-life care
3. individuals incapable of providing informed consent
4. patients who decline participation.

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who were treated in the emergency rescue room
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive score | At the time of inclusion in the study
  The cognitive scores obtained through questionnaire surveys